CLINICAL TRIAL: NCT01045798
Title: MSG-04 (Also Known as Merck Caspofungin Protocol 067): A Pilot, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Caspofungin Empirical Therapy for Invasive Candidiasis in High-Risk Patients in the Critical Care Setting
Brief Title: Pilot Feasibility Study With Patients Who Are at High Risk For Developing Invasive Candidiasis in a Critical Care Setting (MK-0991-067)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low participant enrollment: 15 enrolled of 114 planned
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Mycoses Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0991-067; 2010_502 (Other: Merck)
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Results first posted 2013-05-10 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Invasive Candidiasis
Keywords: Candidiasis; Invasive Candidiasis; Fungal Infection; Empirical Therapy
MeSH Terms: conditions — Candidiasis, Invasive; Candidiasis; Mycoses | interventions — Caspofungin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caspofungin (Experimental): caspofungin acetate
  Interventions: Drug: Caspofungin acetate
- Placebo (Placebo Comparator): normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caspofungin acetate — 70 mg of caspofungin administered intravenously (IV) on Day 1 followed by 50 mg daily for at least 6 additional days (maximum duration study therapy is 14 days)
  Other Names: caspofungin; MK-0991; Cancidas®
  Arms: Caspofungin
Drug: Placebo — Placebo to caspofungin (normal saline) on Day 1 followed by placebo daily for at least 6 additional days (maximum duration study therapy is 14 days)
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
This is a pilot feasibility study that investigates antifungal therapy with caspofungin in patients at high-risk for developing invasive candidiasis in a critical care setting.

DETAILED DESCRIPTION:
Hypothesis: In high-risk non-neutropenic participants in the ICU, the proportion of participants discontinued from study therapy in order to be empirically treated with antifungal therapy for suspected candidiasis outside of the context of this protocol is less than 20% (i.e., the upper bound of the 95% confidence interval for the observed proportion is less than 20%).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for a minimum of 3 days in an ICU and expectation to stay in the ICU for at least another 48 hours
* Meets the following high-risk criteria: Requires mechanical ventilation at the time of study entry; and has a central venous catheter in place at the time of study entry; and is receiving broad spectrum antibiotics at the time of study entry; AND meets at least one of the following criteria: Required parenteral nutrition during the current ICU admission; or required renal dialysis during the current ICU admission; or had major surgery during or within the 7 days before the current ICU admission; or was diagnosed with pancreatitis during or within the 7 days before the current ICU admission; or required systemic steroids or other immunosuppressive agents during or within the 7 days before the current ICU admission
* Meets at least one of the following criteria of suspected infection at the time of study entry or within the 24 hours before study entry: Temperature ≥38° C or ≤36° C (oral equivalent); or hypotension (systolic blood pressure of <90 mm Hg) or significant drop in blood pressure (40 mm Hg) from the participant's normal baseline; or elevated white blood cell count of ≥12,000/mm^3
* Candida is growing in at least one non-sterile culture site collected during the current ICU admission
* Female of childbearing potential has a negative serum or urine pregnancy test before enrollment

Exclusion Criteria:

* Females pregnant or breast feeding
* History of allergy, hypersensitivity, or any serious reaction to caspofungin or another member of the echinocandin class (e.g., micafungin, anidulafungin)
* Neutropenia or expected to develop neutropenia during study therapy
* Diagnosis of acquired immune deficiency syndrome (AIDS), aplastic anemia, or chronic granulomatous disease
* Diagnosis of moderate or severe hepatic insufficiency
* Patient not expected to survive at least 24 hours
* Received systemic (IV or oral) antifungal therapy within 10 days before study entry
* Active diagnosis of proven or probable invasive fungal infection (IFI)
* Currently on or has received an investigational agent within 10 days before study entry
* Any condition or concomitant illness which might confuse the study results or pose additional risk in administering the study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated early due to low participant enrollment.
  One of the 15 participants randomized to treatment inappropriately received a systemic antifungal agent before starting study drug and was not included in the baseline characteristics, safety, or efficacy analyses.
Groups:
- Caspofungin: Caspofungin 70 mg caspofungin administered intravenously (IV) on Day 1 followed by 50 mg daily for at least 6 additional days (maximum duration study therapy is 14 days)
Period: Overall Study
Arm/Group | Caspofungin | Placebo
Started | 6 | 9
Completed | 4 | 5
Not Completed | 2 | 4
Not completed — Changed to Open-Label Caspofungin | 1 | 0
Not completed — Invasive Fungal Infection at Baseline | 0 | 1
Not completed — Changed to Other Antifungal Therapy | 1 | 2
Not completed — Received Systemic Antifungal Prestudy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caspofungin | Placebo | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (20.1) | 53.0 (10.6) | 56.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Discontinued From Study Therapy to be Treated With Empirical Antifungal Therapy Outside of the Context of the Study.
Description: The feasibility of conducting a major randomized study of caspofungin for empirical therapy for invasive candidiasis in high-risk non-neutropenic intensive care unit (ICU) participants was to be assessed by the incidence of study therapy discontinuations due to investigators choosing to treat participants with empirical antifungal therapy outside of the context of this protocol.
  Study drug was administered for a minimum of 7 days to a maximum of 14 days provided participants had no evidence of confirmed breakthrough invasive Candida infection while receiving study drug.
Time Frame: 1 to 14 days
Population: Of the 114 participants anticipated to enroll in this study, 15 actually enrolled and only 14 received study drug. The participant who did not receive study drug was discontinued; the remaining 14 received at least one dose of study drug, met inclusion/exclusion criteria, and therefore qualified for the full analysis set used for summary analyses.
Measure: Number; unit: Participants
Arm/Group | Caspofungin | Placebo
Number analyzed (Participants) | 6 | 8
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: First dose of study drug through up to 14 days post-treatment
Description: All participants who received at least one dose of study drug were included in the safety analyses.
Arm/Group | Caspofungin | Placebo
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/8
Other Adverse Events (participants affected / at risk) | 4/6 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caspofungin (N=6) | Placebo (N=8)
Cardiac arrest (Cardiac disorders) | 1 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 1
Renal abscess (Renal and urinary disorders) | 0 | 1
Pneumonia due to Pseudomonas (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Tracheostomy (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Caspofungin (N=6) | Placebo (N=8)
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Hypoglycaemia (Endocrine disorders) | 0 | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal bleed (Gastrointestinal disorders) | 0 | 1
Medical device complication (General disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatic shock (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Vancomycin-resistant enterococcal infection (Infections and infestations) | 1 | 0
Bilirubin elevated (Investigations) | 1 | 0
Clostridium difficile toxin test positive (Investigations) | 1 | 0
Elevated liver enzymes (Investigations) | 0 | 1
Late diastolic murmur (Investigations) | 1 | 0
Liver enzyme abnormal (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Unresponsive (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchoconstriction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia due to pseudomonas (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin tear (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal aortic aneurysm (Vascular disorders) | 1 | 0
Acute hypotension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
This study was terminated early due to low participant enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.